CLINICAL TRIAL: NCT03870334
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter Study to Evaluate Efficacy and Safety of Oral BT-11 in Moderate to Severe Crohn's Disease
Brief Title: Efficacy and Safety of Oral BT-11 in Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision of Landos Biopharma (not related to safety or efficacy)
Sponsor: NImmune Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BT-11-202
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is a phase 2 randomized, placebo-controlled, double-blind, parallel-group multicenter induction study. The purpose of this study is to evaluate the efficacy and safety of oral BT-11 induction compared to placebo in subjects with moderate to severe CD. Approximately 100 sites will participate from Europe and the USA. A total of 150 subjects with moderate to severe CD (CDAI Score 220-450 and a Simplified Endoscopic Index of Severity of Crohn's Disease (SES-CD) SCORED ≥ 6 (≥ 4 for isolated ileitis) will be randomized in a 1:1 ratio to receive BT-11 1,000 mg or placebo. Each of the treatment arms will comprise 75 subjects. The randomization will be stratified by prior exposure to biologic therapy for CD (yes/no) and corticosteroid use at baseline (yes/no). The study consists of a 28-day screening period, a 12-week induction phase, and a 2-week post-treatment safety follow-up period.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BT-11 880 mg (Experimental): Oral once daily tablet
  Interventions: Drug: BT-11 880 mg
- Placebo (Placebo Comparator): Oral once daily tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BT-11 880 mg — Oral once daily tablet
  Arms: BT-11 880 mg
Drug: Placebo — Oral once daily tablet
  Arms: Placebo

SUMMARY:
This is a phase 2 randomized, placebo-controlled, double-blind, parallel-group multicenter induction study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects aged 18 to 75 years with a diagnosis of CD for at least 3 months;
2. Moderately to severely active CD as defined by: a CDAI score of 220 450, and an SES-CD scored ≥ 6 ( ≥ 4 for isolated ileitis) (centrally read);

Key exclusion criteria:

1. Ulcerative colitis;
2. Known current bacterial or parasitic pathogenic enteric infection; live virus vaccination within 12 weeks of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Study Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BT-11 880 mg | Placebo
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BT-11 880 mg | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.7) | 39.9 (13.7) | 38.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 11 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission Rate
Description: Clinical remission defined by CDAI score <150.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BT-11 880 mg | Placebo
Number analyzed (Participants) | 12 | 11
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | BT-11 880 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 7/12 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BT-11 880 mg (N=12) | Placebo (N=11)
Infections and Infestations (Infections and infestations) | 1 | 3
Other (General disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03870334/Prot_SAP_000.pdf